CLINICAL TRIAL: NCT05674981
Title: To Evaluate the Clinical Efficacy of Probiotic in Patients With DKD
Brief Title: To Evaluate the Beneficial Effect of Probiotics on DKD Patients and the Role of Gut Microbiota Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DKD2022
Record Dates: First submitted 2022-12-19; First posted 2023-01-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic kidney disease; gut microbiota; Probiotic; Lactobacillus reuteri; Lactobacillus rhamnosus
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Randomized Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Subjects received two probiotic sachets per day
  Interventions: Dietary Supplement: Probiotic group
- Placebo group (Placebo Comparator): Subjects received two placebo sachets per day
  Interventions: Other: Placebo group

INTERVENTIONS:
Dietary Supplement: Probiotic group — Two-strain probiotic supplement includes Lactobacillus reuteri ADR-1 (alive) and Lactobacillus rhamnosus GM-020 ( alive).
  Other Names: Test group
  Arms: Probiotic group
Other: Placebo group — Same additives to Probiotic group but replace probiotics with corn starch and Maltodextrin.
  Other Names: Control group
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy of probiotics in the treatment of diabetic kidney disease, this study is designed to explore after consumption of probiotics lactobacillus reuteri ADR-1 and lactobacillus rhamnosus GM-020 composite strain powder sachets for 6 months, whether the improvement of blood sugar, kidney related indicators can further improve the course of diabetic kidney disease. The clinical trial predicted that probiotics can improve diabetic kidney disease by changing the intestinal flora by inhibiting harmful bacteria, reduction of systemic oxidative stress, balance carbohydrate and fat metabolism, further preventing the progress of diabetic kidney disease.

DETAILED DESCRIPTION:
WHO predicts that diabetes will become the seventh leading cause of death in 2030. This disease usually causes complications including hypertension, diabetic kidney disease, neuropathy, skin infection, and a high risk of blindness and so on. It demonstrated that probiotics have beneficial effects on several disorders; these beneficial effects include a reduction in allergic symptoms, a decrease in serum cholesterol levels, the prevention of obesity, and an improvement of the digestive system. In recent years, many studies have pointed out that Lactobacillus affects the progression of diabetes kidney disease by controlling blood sugar. From 2017 to 2020, 8 clinical trials conducted related research to explore the clinical benefits of probiotics on diabetic kidney disease. It was found that the indicators related to kidney function have ameliorated significantly, including improving glomerular function, blood sugar control, insulin metabolism, inflammatory substances in serum, and even oxidative stress factors, etc.

In a previous study, Lactobacillus strain ADR-1 was selected to verify the efficacy by utilizing HFD (High-fructose-fed) rats model, the result shows reductions in serum HbA1c and liver injury after oral gavage for 14 weeks. Afterward, a double-blind, randomized, placebo-group human clinical trial was conducted, recruiting 68 subjects with type 2 diabetes to evaluate the intestinal flora and blood sugar-related indicators, among which the metabolic indicators had significant changes. After taking it for 3 and 6 months, HbA1c and cholesterol were significantly reduced compared to the Placebo group, it was also found that the L.reuteri flora had a significant increase in the intestinal flora while the same pattern was found in the Bifidobacterium flora accordingly. This result represents the development of a positive correlation between Lactobacillus and Bifidobacterium for the intestinal flora. Furthermore, GM-020 has been proved by mouse model experiments to slow down kidney diseases, including the improvement of related indicators of renal function, serum urea nitrogen (BUN), and creatinine (Creatinine), and it shows dose-dependent variation. The combination of these two strains of probiotics is predicted to improve the metabolical index of diabetic kidney disease.

This clinical trial will explore the health-promoting effect of probiotics on patients with diabetic kidney disease, and fully explore how probiotics can improve the good bacteria and reduce the bad bacteria by changing the intestinal flora to achieve anti-inflammatory effects, Chronic inflammation, reduce systemic oxidative stress, balances carbohydrate and fat metabolism, and prevents the progression of diabetic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 80 years old
* Suffering from type 2 diabetes and stable medication for 3 months
* Detection of HbA1c before meals between 7% and 10%
* Stage 1-3a diabetic nephropathies (eGFR > 45 mL/min)
* Microalbuminuria estimated between 30 to 300 mg/day

Exclusion Criteria:

* Patients with Type I Diabetes Mellitus
* Patients with inflammatory bowel disease, liver disease, liver cirrhosis, systemic lupus erythematosus, malignancy, and high blood pressure.
* Patients with hypoglycemic coma, Diabetic ketoacidosis, hyperosmolar non-ketotic diabetic coma, or diabetes mellitus acute complications.
* Acute infection medical history in past 3 month
* Fasting blood glucose >13.3 mmol/L
* GPT>100U/L (2.5 times than usual situation)
* Vulnerable population (Including breeding or pregnant women, prisoner, aboriginal, disabled population)
* Smoker or Alcoholic
* Taking Antibiotics in past 1 month
* Stably taking probiotics supplements in past 1 months (Yogurt or dairy products were excluded)
* Taking immunosuppressive drug, angiotensin-converting enzyme inhibitors, or angiotensin receptor blockers in past 3 months

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Cys-C (Cystatin C) level at 3 months | 3 months
  Blood samples will be collected to examine the variation of Cys-C (Cystatin C) from baseline at 3 months.
Change from baseline in Cys-C (Cystatin C) level at 6 months | 6 months
  Blood samples will be collected to examine the variation of Cys-C from baseline at 6 months.

SECONDARY OUTCOMES:
Change from baseline in BMI (Body Mass Index) at 3 months | 3 months
  BMI will be calculated with weight and height combined in kg/m^2.
Change from baseline in BMI (Body Mass Index) at 6 months | 6 months
  BMI will be calculated with weight and height combined in kg/m^2.
Change from baseline in Waist and hip circumference at 3 months | 3 months
  Waist and hip circumference will take down in centimeters.
Change from baseline in Waist and hip circumference at 6 months | 6 months
  Waist and hip circumference will take down in centimeters.
Change from baseline in blood pressure at 3 months | 3 months
  The unit of measurement of blood pressure is mmHg. Both systolic and diastolic blood pressure will be measured.
Change from baseline in blood pressure at 6 months | 6 months
  The unit of measurement of blood pressure is mmHg. Both systolic and diastolic blood pressure will be measured.
Change from baseline in levels of FPG (Fasting Plasma Glucose) at 3-months | 3 months
  Fasting blood samples will be collected to examine variation in FPG in uIU/mL.
Change from baseline in levels of FPG at 6-months | 6 months
  Fasting blood samples will be collected to examine variation in FPG in uIU/mL.
Change from baseline in levels of serum insulin at 3-months | 3 months
  Fasting blood samples will be collected to examine variation in serum insulin in uIU/mL.
Change from baseline in levels of serum insulin at 6-months | 6 months
  Fasting blood samples will be collected to examine variation in serum insulin in uIU/mL.
Change from baseline in levels of HbA1c (Hemoglobin A1C) at 3-months | 3 months
  Fasting blood samples will be collected to investigate the levels of HbA1c in %.
Change from baseline in levels of HbA1c at 6-months | 6 months
  Fasting blood samples will be collected to investigate the levels of HbA1c in %.
Change from baseline in levels of HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) at 3-months | 3 months
  The equation of HOMA-IR=(insulin (mIU/L) and glucose (mg/dL))/405)
Change from baseline in levels of HOMA-IR at 6-months | 6 months
  The equation of HOMA-IR=(insulin (mIU/L) and glucose (mg/dl))/405)
Change from baseline in levels of HOMA-β (Homeostatic Model Assessment for β-cell function) at 3-months | 3 months
  The equation of HOMA-β=20 × fasting insulin (μIU/ml)/fasting glucose (mmol/ml) - 3.5
Change from baseline in levels of HOMA-β (Homeostatic Model Assessment for β-cell function) at 6-months | 6 months
  The equation of HOMA-β=20 × fasting insulin (μIU/ml)/fasting glucose (mmol/ml) - 3.5
Change from baseline in levels of QUICKI (Quantitative Insulin Sensitivity Check Index) at 3-months | 3 months
  The equation of QUICKI=1 / [log(Fasting Insulin (µU/ml) + log(Fasting Glucose (mg/dL))]
Change from baseline in levels of QUICKI (Quantitative Insulin Sensitivity Check Index) at 6-months | 6 months
  The equation of QUICKI=1 / [log(Fasting Insulin (µU/ml) + log(Fasting Glucose (mg/dL))]
Change from baseline in the level of GA (Glycated albumin) at 3-months | 3 months
  Blood samples will be collected to examine changes in GA in mg/dL.
Change from baseline in the level of GA (Glycated albumin) at 6-months | 6 months
  Blood samples will be collected to examine changes in GA in mg/dL.
Change from baseline in the level of CRE (Creatinine) at 3-months | 3 months
  Blood samples will be collected to examine changes in CRE in mg/dL.
Change from baseline in the level of CRE at 6-months | 6 months
  Blood samples will be collected to examine changes in CRE in mg/dL.
Change from baseline in the level of BUN (Blood Urea Nitrogen) at 3-months | 3 months
  Blood samples will be collected to examine changes in BUN in mg/dL.
Change from baseline in the level of BUN at 6-months | 6 months
  Blood samples will be collected to examine changes in BUN in mg/dL.
Change from baseline in the level of K+ (Potassium) at 3-months | 3 months
  Blood samples will be collected to examine changes from baseline in K+ in mg/dL.
Change from baseline in the level of K+ at 6-months | 6 months
  Blood samples will be collected to examine changes from baseline in K+ in mg/dL.
Change from baseline in the level of Urine protein/albumin at 3-months | 3 months
  Urine samples will be collected to examine changes in Urine protein/albumin in mg/dL.
Change from baseline in the level of Urine protein/albumin at 6-months | 6 months
  Urine samples will be collected to examine changes in Urine protein/albumin in mg/dL.
Change from baseline in the level of Urine microalbuminuria/creatinine at 3-months | 3 months
  Urine samples will be collected to examine changes from baseline in Urine protein/albumin in mg/dL.
Change from baseline in the level of Urine microalbuminuria/creatinine at 6-months | 6 months
  Urine samples will be collected to examine changes from baseline in Urine protein/albumin in mg/dL.
Change from baseline in the level of Urine acid at 3-months | 3 months
  Urine samples will be collected to examine changes in Urine protein/albumin in mg/dL.
Change from baseline in the level of Urine acid at 6-months | 6 months
  Urine samples will be collected to examine changes in Urine protein/albumin in mg/dL.
Change from baseline in the level of CG (The Cockcroft and Gault formula) at 3-months | 3 months
  CG will be calculated with creatinine, age, weight, gender. The equation of CG = (((140 - age in years) x (weight in kg)) x 1.23) / (serum creatinine in micromol/l).
Change from baseline in the level of CG at 6-months | 6 months
  CG will be calculated with creatinine, age, weight, gender. The equation of CG = (((140 - age in years) x (weight in kg)) x 1.23) / (serum creatinine in micromol/l).
Change from baseline in the level of eGFR (Estimated Glomerular Filtration Rate) at 3-months | 3 months
  eGFR will be estimated according to the CKD-EPI Creatinine Equation (2021) which is calculated with serum creatinine, Cystatin C, age, gender.
Change from baseline in the level of eGFR (Estimated Glomerular Filtration Rate) at 6-months | 6 months
  eGFR will be estimated according to the CKD-EPI Creatinine Equation (2021) which is calculated with serum creatinine, Cystatin C, age, gender.
Change from baseline in levels of blood lipid-related Index at 3 months | 3 months
  Blood samples will be collected to examine variation in TG (Triglyceride), TC (Total Cholesterol), VLDL (Very-Low-Density Lipoprotein), LDL (Low-density lipoprotein), HDL (High-density lipoprotein).
Change from baseline in levels of blood lipid-related Index at 6 months | 6 months
  Blood samples will be collected to examine variation in TG (Triglyceride), TC (Total Cholesterol), VLDL (Very-Low-Density Lipoprotein), LDL (Low-density lipoprotein), HDL (High-density lipoprotein).
Change from baseline in levels of cytokines Index at 3 months | 3 months
  Blood samples will be collected to examine variation in hs-CRP (high-sensitivity C-reactive protein), IL-6 (Interleukin-6), IL-18 (Interleukin-18), IL -1-α (Interleukin-1-α), IL-1β (Interleukin-1 β), TNF-α (Tumor necrosis factor-α), NGAL (Neutrophil Gelatinase-Associated Lipocalin), sTNFR1 (Soluble tumour necrosis factor receptor-1), PGRN (Progranulin). All the indexes will be recorded in in pg/mL.
Change from baseline in levels of cytokines Index at 6 months | 6 months
  Blood samples will be collected to examine variation in hs-CRP, IL-6, IL-18, IL-1-α, IL-1β, TNF-α, NGAL, sTNFR1, PGRN. All the indexes will be recorded in in pg/mL.
Change from baseline in levels of TIBC (Total Iron-Binding Capacity) at 3-months | 3 months
  TIBC will be calculated by summing the values of serum iron and UIBC(unsaturated iron-binding capacity) which is examed from blood samples.
Change from baseline in levels of TIBC at 6-months | 6 months
  TIBC will be calculated by summing the values of serum iron and UIBC which is examed from blood samples.
Change from baseline in the level of SCFA (Short Chain Fatty Acids) at 6 months | 6 months
  Stool samples will be collected to examine variation in SCFA (Short Chain Fatty Acids).
Change from baseline in the level of TMAO (Trimethylamine N-oxide) at 3-months | 3 months
  Blood samples will be collected to examine variation in TMAO in μmol/L.
Change from baseline in the level of TMAO at 6-months | 6 months
  Blood samples will be collected to examine variation in TMAO in μmol/L.
Change from baseline in self-record of the International physical activity questionary (IPAQ) in physical assessment at 6 months | 6 months
  The questionnaire will be recorded the laborious activity by the subject himself/herself before and after the treatment.
Change from baseline in gut microbiota at 6 months | 6 months
  The analysis of Gut microbiota will utilize DNA sequencing to investigate the intestinal microbiota through stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Sun Yang, PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan, Taiwan